CLINICAL TRIAL: NCT05967689
Title: An Open-Label, Phase 2b, Global Multicenter Cohort Trial to Assess the Safety and Efficacy of Zipalertinib in Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer With Exon 20 Insertion and Uncommon/Single or Compound Epidermal Growth Factor Receptor Mutations.
Brief Title: A Study of Zipalertinib in Patients With Advanced Non-Small Cell Lung Cancer With Epidermal Growth Factor Receptor (EGFR) Exon 20 Insertions or Other Uncommon Mutation.
Acronym: REZILIENT2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAS6417-201; 2023-503865-48 (EudraCT Number)
Record Dates: First submitted 2023-07-11; First posted 2023-08-01 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Advanced or Metastatic NSCLC Harboring Epidermal Growth Factor Receptor (EGFR) Exon 20 Insertion (ex20ins) Mutations
Keywords: NSCLC; Carcinoma; Non-Small Cell Lung; Lung disease; locally advanced/ metastatic; ex20ins mutation; Insertion Mutations; EGFR uncommon/ single mutation Phase 2, Phase 2b, Phase II Exon 20; TAS6417/ CLN-081
MeSH Terms: conditions — Carcinoma; Lung Diseases | interventions — zipalertinib

STUDY DESIGN:
Intervention Model Description: 6 Cohorts based on eligibility criteria
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- Cohort A ("prior ex20ins treatment") (Experimental): Cohort A ("prior ex20ins treatment") participants will receive zipalertinib orally twice a day (BID) continuously until documentation of progressive disease (PD) or until other withdrawal criteria are met, whichever comes first.
  Interventions: Drug: TAS6417
- Cohort B ("first-line treatment") (Experimental): Cohort B participants will receive zipalertinib orally, BID continuously until documentation of PD or until other withdrawal criteria are met, whichever comes first.
  Interventions: Drug: TAS6417
- Cohort C ("active brain mets") (Experimental): Cohort C participants will receive zipalertinib orally, BID continuously until documentation of PD or until other withdrawal criteria are met, whichever comes first.
  Interventions: Drug: TAS6417
- Cohort D ("other uncommon EGFRmts"). (Experimental): Cohort D participants will receive zipalertinib orally, BID continuously until documentation of PD or until other withdrawal criteria are met, whichever comes first.
  Interventions: Drug: TAS6417
- DDI Substudy: CYP Cocktail Group (Experimental): Participants will receive a single dose of CYP enzyme probe substrates (CYP cocktail) alone prior to the start of zipalertinib dosing and a single dose of CYP cocktail in combination with zipalertinib at steady state. Zipalertinib will be dosed, orally BID in Cycle 1 (cycle length = 21 days), followed by continuous treatment with zipalertinib until documentation of PD or until other withdrawal criteria are met, whichever comes first.
  Interventions: Drug: TAS6417; Drug: CYP Cocktail
- DDI Substudy: Transporter Cocktail Group (Experimental): Participants will receive a single dose of transporter probe substrates (Transporter cocktail) alone prior to the start of zipalertinib dosing and a single dose of Transporter cocktail in combination with zipalertinib at steady state. Zipalertinib will be dosed, orally BID in Cycle 1 (cycle length = 21 days), followed by continuous treatment with zipalertinib until documentation of PD or until other withdrawal criteria are met, whichever comes first.
  Interventions: Drug: TAS6417; Drug: Transporter Cocktail
- Dose Optimization Substudy: Arm A (Experimental): Participants will receive zipalertinib, orally, at Arm A dose, BID, continuously in 21-day treatment cycles until the participant meets any of the treatment discontinuation criteria.
  Interventions: Drug: TAS6417
- Dose Optimization Substudy: Arm B (Experimental): Participants will receive zipalertinib, orally, at Arm B dose, BID, continuously in 21-day treatment cycles until the participant meets any of the treatment discontinuation criteria.
  Interventions: Drug: TAS6417

INTERVENTIONS:
Drug: TAS6417 — Oral tablets
  Other Names: CLN-081; zipalertinib
Drug: CYP Cocktail — Single dose of CYP enzyme probe substrates (CYP cocktail) alone prior to the start of zipalertinib dosing and a single dose of CYP cocktail in combination with zipalertinib at steady state.
  Arms: DDI Substudy: CYP Cocktail Group
Drug: Transporter Cocktail — Single dose of transporter probe substrates (Transporter cocktail) alone prior to the start of zipalertinib dosing and a single dose of Transporter cocktail in combination with zipalertinib at steady state.
  Arms: DDI Substudy: Transporter Cocktail Group

SUMMARY:
The purpose of this study is to evaluate the safety, efficacy and pharmacokinetics (PK) of zipalertinib in participants with locally advanced or metastatic Non-Small Cell Lung Cancer (NSCLC) harboring EGFR ex20ins mutations and other mutations.

DETAILED DESCRIPTION:
This study will evaluate the safety and efficacy of zipalertinib in participants with locally advanced or metastatic NSCLC harboring EGFR ex20ins mutations or other uncommon/single or compound Epidermal Growth Factor Receptor Proteins Mutations (EGFRmts). The drug-drug interaction (DDI) substudy will assess the potential DDI effects of zipalertinib on the pharmacokinetics (PK) of cytochrome P450 (CYP) enzyme substrates and transporter substrates and also evaluate the relationship between zipalertinib concentration and QT interval change from baseline. Additionally, dose optimization substudy will be conducted to confirm an optimized dose of zipalertinib monotherapy.

Participants will be enrolled into 1 of the 4 following cohorts:

* Cohort A ("prior ex20ins treatment") will include participants harboring EGFR ex20ins who have progressed on or after initial treatment with standard platinum-based chemotherapy and prior treatment with an ex20ins agent for their advanced disease (administered together or separately).
* Cohort B ("first-line") will include participants harboring EGFR ex20ins who have not received prior treatment for advanced or metastatic disease and are not appropriate candidates for first-line doublet platinum-based chemotherapy or have refused first-line doublet platinum-based chemotherapy.
* Cohort C ("active brain mets") will include participants harboring EGFR ex20ins or other uncommon single or compound EGFRmts and active brain metastases and/or leptomeningeal disease (LMD). Participants may or may not have had prior treatment for advanced disease.
* Cohort D ("other uncommon EGFRmts") will include participants harboring other non-ex20ins, excluding C797S (uncommon single or compound) EGFRmts who have not received prior systemic therapy for their locally advanced or metastatic NSCLC disease.

For DDI substudy, participants will be enrolled in two groups:

* CYP Cocktail Group will receive a single dose of cocktail of CYP enzyme probe substrates (CYP cocktail) alone prior to the start of zipalertinib dosing and a single dose of CYP cocktail in combination with zipalertinib at steady state.
* Transporter Cocktail Group will receive a single dose of transporter probe substrates (Transporter cocktail) alone prior to the start of zipalertinib dosing and a single dose of Transporter cocktail in combination with zipalertinib at steady state.

For dose-optimization substudy, participants with locally advanced or metastatic NSCLC harboring epidermal growth factor receptor protein ex20ins mutations (EGFRmts) will be randomized to receive zipalertinib at different doses with continuous daily dosing until any discontinuation criterion is met. Participants will be enrolled into two groups: Arm A and Arm B, in which they will receive different doses of zipalertinib.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. ≥18 years of age (or meets the country's regulatory definition of legal adult age, whichever is greater.
3. Pathologically confirmed, locally advanced or metastatic NSCLC meeting all the following criteria:

   Cohort A participants:
   * Documented EGFR ex20ins status, as determined by local testing performed at a Clinical Laboratory Improvement Amendments (CLIA) certified (United States [US]) or locally certified laboratory (outside the US).
   * Progressed on or after systemic therapy with an agent targeting ex20ins, either alone or in combination with standard platinum-based chemotherapy for the treatment of advanced disease. Participants who discontinued previous treatment due to unacceptable toxicity are eligible.

     i. Permitted prior ex20ins therapies include: amivantamab, sunvozertinib (DZD9008), and BLU451. Other prior ex20ins--directed treatment may be discussed with the Sponsor for eligibility assessment.
   * Participants with brain metastasis must be neurologically stable. Participants must have received central nervous system (CNS)-directed therapy and have no evidence of progression for at least 4 weeks after CNS-directed treatment, as ascertained by clinical examination and brain imaging (magnetic resonance imaging [MRI] or computed tomography [CT] scan) during the Screening Period. Additionally, they must be on a stable or decreasing dose of corticosteroids and/or anti-convulsant medications for at least 2 weeks prior to the first dose of study treatment. Participants with a history of uncontrolled seizures or LMD are not eligible.

   Cohort B participants:
   * Documented EGFR ex20instatus, as determined by local testing performed at a CLIA-certified (US) or locally certified laboratory (outside the US).
   * Participants who have not received prior treatment for advanced or metastatic disease and who are not appropriate candidates for first-line doublet platinum-based chemotherapy based on Investigator judgment or has refused first-line doublet platinum-based chemotherapy following discussion with the Investigator. Prior adjuvant/neoadjuvant treatment for early-stage disease must have been completed >6 months prior to the first dose of study treatment.
   * Participants with brain metastasis must be neurologically stable. Participants must have received CNS-directed therapy and have no evidence of progression for at least 4 weeks after CNS-directed treatment, as ascertained by clinical examination and brain imaging (MRI or CT scan) during the Screening Period, and they must be on a stable or decreasing dose of corticosteroids and/or anti-convulsant medications for at least 2 weeks prior to the first dose of study treatment. Participants with history of uncontrolled seizures or LMD are not eligible.

   Cohort C participants:
   * Documented ex20ins or other uncommon single or compound EGFR non-ex20ins status, as determined by local testing performed at a CLIA-certified (US) or locally certified laboratory (outside the US).
   * Presence of brain metastasis(es) characterized as at least one of the following:

     * Newly diagnosed and/or progressive brain metastasis(es) measurable by Response Assessment in Neuro-oncology Brain Metastases (RANO-BM) criteria and not subjected to CNS-directed therapy, AND/OR
     * LMD measurable or non-measurable by RANO-BM criteria and confirmed by a positive cerebrospinal fluid cytology, or unequivocal radiographic and/or clinical determination.
   * Participants may not require other immediate CNS-directed therapy or will likely require other CNS directed anti-tumor therapy during the first cycle of study treatment, as judged by the Investigator.

   Cohort D participants:
   * Documented other uncommon single or compound EGFR non-ex20ins status (excluding C797S), as determined by local testing performed at a CLIA certified (US) or locally certified laboratory (outside the US). A list of eligible mutations will be provided in a separate document.
   * Participants with brain metastasis must be neurologically stable. Participants must have received CNS-directed therapy and have no evidence of progression for at least 4 weeks after CNS- directed treatment, as ascertained by clinical examination and brain imaging (MRI or CT scan) during the Screening Period, and they must be on a stable or decreasing dose of corticosteroids and/or anti-convulsant medications for at least 2 weeks prior to the first dose of study treatment. Participants with history of uncontrolled seizures or LMD are not eligible.
   * Participants who have not received prior systemic therapy for their locally advanced or metastatic NSCLC disease.
   * Prior adjuvant/neoadjuvant treatment for early-stage disease must have been completed >6 months prior to the first dose of study treatment. Participants may not have received prior adjuvant/neoadjuvant treatment with any EGFR tyrosine kinase inhibitor (TKI).
4. Measurable disease per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1).
5. Archival tumor tissue available for submission, with minimum quantity sufficient to evaluate EGFRmt status and, where possible, other biomarkers (details provided in a laboratory manual). Participants with insufficient tissue may be eligible following discussion with the Sponsor.
6. Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0 or 17.
7. Adequate organ function, as defined by the hematologic, renal and hepatic laboratory values.
8. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test prior to administration of the first dose of study treatment. Female participants are not considered to be of childbearing potential if they are post-menopausal (no menses for 12 months without an alternative medical cause) or permanently sterile (hysterectomy, bilateral salpingectomy, or bilateral oophorectomy).
9. Both males and females of reproductive potential must agree to use effective birth control during the study prior to the first dose of study drug and for 1 month after the last dose of study treatment.

DDI Substudy:

1. Participant has pathologically confirmed, locally advanced or metastatic NSCLC:

   a. Documented EGFRmt status as determined by local testing performed at a clinical laboratory improvement amendments (CLIA) certified (US) or locally certified laboratory (outside of the US) local laboratory, defined as either one of the following EGFRmts:
   * ex20ins EGFRmt OR
   * other uncommon, non-ex20ins EGFRmt (eg, G719X, L861Q, or S768I) OR
   * common EGFRmt (eg, ex19del or L858R)
2. Participant has progressed on or after receiving prior standard of care (SoC) systemic therapy for their locally advanced or metastatic NSCLC disease unless:

   * Participant for whom no approved therapy with demonstrated clinical benefit is indicated or available,
   * Participant is intolerant to the available first-line (1L) SoC treatment options, OR
   * Participant has refused 1L SoC treatment options (after being appropriately informed of the treatment options, risks, and benefits).
3. Participants with brain metastasis are eligible if they fulfill all of the criteria below:

   * Have received CNS-directed therapy and have no evidence of progression for at least 4 weeks after CNS- directed treatment, as ascertained by brain imaging (MRI or CT scan) during the Screening Period,
   * Are on a stable or decreasing dose of corticosteroids and/or anti-convulsant medications for at least 2 weeks prior to the first dose of study treatment,
   * Are neurologically stable with no history of uncontrolled seizures.
4. ECOG PS of 0 or 1.

Dose Optimization Substudy:

1. Has pathologically confirmed, locally advanced or metastatic NSCLC meeting all the following criteria:

   1. Documented EGFR ex20ins status, as determined by local testing performed at a CLIA certified (US) or locally certified laboratory (outside the US)
   2. Progressed on or after systemic therapy standard platinum-based chemotherapy for the treatment of advanced disease. Participants who discontinued previous treatment due to unacceptable toxicity are eligible.

   Note: Progression on or after systemic therapy with amivantamab is permitted (eg, given as monotherapy or in combination with chemotherapy).
2. Participants with CNS metastases are eligible if both of the following criteria are met:

   i. Measurable lesions according to RANO-BM defined as a contrast-enhancing lesion that can be accurately measured in at least one dimension, with a minimum size of 10 millimeters (mm), or at least 5 mm if MRI slice thickness is ≤ 1.5 mm ii. Previously received definitive local treatment and have stable CNS disease (defined as being neurologically stable and off corticosteroid for at least 2 weeks prior to enrollment) OR Asymptomatic CNS metastases ≤ 2 cm in size if, in the opinion of the investigator, immediate definitive treatment is not indicated.
3. Measurable disease per RECIST 1.1.
4. Has archival tumor tissue available for submission, with minimum quantity sufficient to evaluate EGFRmt status and, where possible, other biomarkers
5. ECOG PS of 0 or 1.
6. Has adequate organ function.

Exclusion Criteria:

1. Participant is currently receiving an investigational drug in a clinical trial or participating in any other type of medical research judged to be scientifically or medically incompatible with this study.
2. Has received any of the following within the specific time frame specified:

   1. Participant has received Zipalertinib (TAS6417/CLN081) at any time
   2. CNS radiotherapy (gamma knife radiotherapy is allowed) ≤ 12 weeks, thoracic radiotherapy ≤ 28 days, or other palliative radiation ≤ 14 days prior to the first dose of study
   3. Anticancer immunotherapy ≤28 days prior to the first dose of study treatment
   4. Major surgery (excluding placement of vascular access) ≤28 days prior to the first dose of study treatment.
   5. Any prior treatment with an EGFR exon20ins- targeted TKI
   6. Participants with leptomeningeal CNS disease.
3. Have any unresolved toxicity of Grade ≥2 from previous anticancer treatment, except for Grade 2 alopecia or skin pigmentation. Participants with other chronic but stable Grade 2 toxicities may be allowed to enroll after agreement between the Investigator and Sponsor.
4. Past medical history of interstitial lung disease, treatment-related pneumonitis (any grade), or evidence of clinically active interstitial lung disease.
5. Impaired cardiac function or clinically significant cardiac disease including any of the following:

   1. History of congestive heart failure (CHF) Class III/IV according to the New York Heart Association (NYHA) Functional Classification.
   2. Serious cardiac arrhythmias requiring treatment.
   3. Resting corrected QT interval (QTc) >470 msec using Fridericia's formula (QTcF).
6. Is unable to swallow tablets or has any disease or condition that may significantly affect gastrointestinal absorption of zipalertinib (eg, inflammatory bowel disease, malabsorption syndrome, or prior gastric/bowel resection).
7. History of another primary malignancy ≤2 years prior to the date of first dose of study treatment unless at least one of the following criteria are met:

   1. Adequately treated basal or squamous cell carcinoma of the skin
   2. Cancer in situ of the breast or cervix
   3. Participants with previously treated malignancy if all treatment for that malignancy was completed at least 2 years prior to first dose and no evidence of disease
   4. Participants with concurrent malignancy clinically stable and not requiring tumor-directed treatment
8. Known history of hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) that is not controlled with treatment.
9. History of Coronavirus disease 2019 (COVID-19) infection within 4 weeks prior to enrollment and/or has persistent clinically significant pulmonary symptoms related to prior COVID-19 infection.
10. Active bleeding disorders.
11. Known hypersensitivity to the ingredients in zipalertinib or any drugs similar in structure or class.
12. Is pregnant, lactating, or planning to become pregnant.
13. The participant is, in the Investigator's opinion, unable or unwilling to comply with the trial procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2023-07-31 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Cohorts 1-4: Objective Response Rate (ORR) | Up to approximately 2 years
Dose Optimization Substudy: ORR as Assessed by Blinded Independent Central Review (BICR) | Up to approximately 2 years

SECONDARY OUTCOMES:
Cohorts 1-4: Number of Participants With Treatment Emergent Adverse Events (TEAEs) Graded According to the National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE v5.0) | Up to approximately 2 years
Cohorts 1-4: Number of Participants with Clinically Significant Changes in Clinical Laboratory Parameters | Up to approximately 2 years
Cohorts 1-4: Number of Participants with Clinically Significant Changes in Vital Signs | Up to approximately 2 years
Cohorts 1-4: Number of Participants with Clinically Significant Changes in Electrocardiogram (ECG) Parameters | Up to approximately 2 years
Cohorts 1-4: Number of participants With Change in Left Ventricular Ejection Fraction (LVEF) Evaluated Using Electrocardiography (ECHO) and Multigated Acquisition (MUGA) Scan | Up to approximately 2 years
Cohorts 1-4: Disease Control Rate (DCR) | Up to approximately 2 years
Cohorts 1-4: Duration of Response (DoR) | Up to approximately 2 years
Cohorts 1-4: Progression-free Survival (PFS) | Up to approximately 2 years
Cohorts 1-4: Overall Survival (OS) | Up to approximately 2 years
Cohort C: Intracranial (i) Overall Response Rate (iORR) | Up to approximately 2 years
Cohort C: Intracranial Duration of Complete Response (iDCR) | Up to approximately 2 years
Cohort C: Intracranial Duration of Response (iDoR) | Up to approximately 2 years
Cohorts 1-4: Minimum Plasma Concentration (Cmin) of Zipalertinib | Up to approximately 2 years
DDI Substudy: Change From Baseline in QT interval Corrected for Heart Rate using Fridericia's formula (QTcF) Interval Following Zipalertinib Administration in CYP Cocktail Group | Cycle 1 (cycle length = 21 days)
DDI Substudy: Geometric Mean Maximum Plasma Concentration (Cmax) After Multiple Dose Administration of Zipalertinib in CYP Group and Transporter Cocktail Groups | Cycle 1 (cycle length = 21 days)
DDI Substudy: Geometric Mean Area Under Curve (AUC) After Multiple Dose Administration of Zipalertinib in CYP Group and Transporter Cocktail Groups | Cycle 1 (cycle length = 21 days)
DDI Substudy: Number of Participants with Treatment-Emergent Adverse Events (TEAEs) in CYP Group and Transporter Cocktail | Cycle 1 (cycle length = 21 days)
Dose Optimization Substudy: Duration of Response (DoR) as Assessed by BICR and Investigator | Up to approximately 2 years
Dose Optimization Substudy: Time to Response as Assessed by BICR and Investigator | Up to approximately 2 years
Dose Optimization Substudy: Percent Change in Tumor Size From Baseline as Assessed by BICR and Investigator | Up to approximately 2 years
Dose Optimization Substudy: DCR as Assessed by BICR and Investigator | Up to approximately 2 years
Dose Optimization Substudy: PFS as Assessed by BICR and Investigator | Up to approximately 2 years
Dose Optimization Substudy: 6 Month PFS Rate | Up to approximately 2 years
Dose Optimization Substudy: ORR as Assessed by Investigator | Up to approximately 2 years
Dose Optimization Substudy: Overall Survival (OS) | Up to approximately 2 years
Dose Optimization Substudy: Intracranial ORR (iORR) per Response Assessment in Neuro-oncology Brain Metastases (RANO-BM) Criteria | Up to approximately 2 years
Dose Optimization Substudy: Intracranial Duration of Response (iDOR) | Up to approximately 2 years
Dose Optimization Substudy: Intracranial Disease Control Rate (iDCR) | Up to approximately 2 years
Dose Optimization Substudy: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to approximately 2 years

CONTACTS AND LOCATIONS:
Locations (80):
- United States (18):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - City of Hope - Duarte, Duarte, California
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Memorial Sloan Kettering Cancer Center - Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center - Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Cancer Center - Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center - Commack, Commack, New York
  - Memorial Sloan Kettering Cancer Center - Westchester, Harrison, New York
  - MSK Cancer Center, Long Island City, New York
  - Memorial Sloan Kettering Cancer Center - Nassau, Uniondale, New York
  - Gabrail Cancer and Research Center, Canton, Ohio
  - Zangmeister Cancer Center, Columbus, Ohio
  - The Toledo Clinic Cancer Center, Toledo, Ohio
  - SCRI Oncology Partners, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Virginia Cancer Specilalist, Fairfax, Virginia
  - IDS Pharmacy, Milwaukee, Wisconsin
- Australia (3):
  - Bankstown-Lidcombe Hospital, Bankstown, New South Wales
  - Genesis Care North Shore, Saint Leonards, New South Wales
  - Joondalup Hospital Pharmacy, Joondalup, Western Australia
- William Osler Health System - Brampton Civic Hospital, Brampton, Canada
- France (9):
  - Nouvel Hôpital Civil, Strasbourg, Aslace
  - Centre Leon Berard, Lyon, Auvergne-Rhône-Alpes
  - CHU Caen Normandie, Caen, Basse-Normandie
  - Centre Hospitalier Universitaire Limoges, Limoges, Limousin
  - Hopital Haut Leveque, Pessac, Nouvelle-Aquitaine
  - Hôpital Nord Marseille, Marseille, Provence-Alpes-Côte d'Azur Region
  - Hopital Nord Laennec, Saint-Herblain
  - Hopital Ambroise Pare, Boulogne-Billancourt, Île-de-France Region
  - Institut Curie, Paris, Île-de-France Region
- Germany (4):
  - Gesundheit Nordhessen Holding AG, Kassel, Hassen
  - Uniklinik Dresden, Dresden
  - UKGM Studienzentrale, Giessen
  - UKR Innere Med II Pneumologie, Regensburg
- Queen Mary Hospital, Pok Fu Lam, Hong Kong Island, Hong Kong
- Italy (6):
  - Azienda Ospedaliero - Universitaria Careggi, Florence, Florence
  - Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori" - IRST, Meldola, Forli-Cesena
  - Azienda Socio-Sanitaria Territoriale di Cremona, Cremona
  - Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS) - Ospedale San Raffaele, Milan
  - Azienda Ospedaliero-Universitaria di Parma, Parma
  - Ospedale S. Maria delle Croci, Ravenna
- Japan (10):
  - Aichi Cancer Center, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - NHO Kyushu Cancer Center, Fukuoka, Hukuoka
  - Sendai Kousei Hospital, Sendai, Miyagi
  - Niigata Cancer Center Hospital, Niigata, Niigata
  - Kindai University Hospital, Sayama, Osaka
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka
  - National Cancer Center Hospital, Chuo Ku, Tokyo
  - Cancer Institute Hospital of JFCR, Koto-ku, Tokyo
  - Okayama University Hospital, Okayama
- South Korea (10):
  - National Cancer Center - Korea, Goyang-si, Gyeonggi-do
  - Saint Vincent's Hospital, Suwon, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Gyeongsang National University Hospital, Jinju, Gyeongsangnamdo [Kyongsangnam-do]
  - Inha University Hospital, Incheon, Incheon Gwang'yeogsi [Inch'on-Kwangyokshi]
  - Chonnam National University Hwasun Hospital, Hwasun-gun, Jeollanam-do
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi [Seoul-T'ukpyolshi]
  - Asan Medical Center, Seoul, Seoul Teugbyeolsi [Seoul-T'ukpyolshi]
  - Korea University Guro Hospital, Seoul, Seoul Teugbyeolsi [Seoul-T'ukpyolshi]
  - Seoul St. Mary's Hospital, Soeul, Seoul Teugbyeolsi [Seoul-T'ukpyolshi]
- Spain (9):
  - Hospital Regional Universitario de Málaga - Hospital General, Málaga, Malaga
  - UOMi Clinica Mi Tres Torres, Barcelona
  - Hospital Quirónsalud Barcelona, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Complejo Hospitalario de Jaen, Jaén
  - MD Anderson Cancer Center Madrid, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital La Paz, Madrid
- Turkey (Türkiye) (5):
  - Istinye Üniversite Hastanesi Liv Hospital Bahcesehir, Esenyurt, Istanbul
  - Medical Park Seyhan Hastanesi, Adana
  - Trakya Üniversitesi Saglik Arastirma ve Uygulama Merkezi, Edirne
  - Bagcilar Medipol Mega Universite Hastanesi, Istanbul
  - Prof. Dr. Suleyman Yalcin Sehir Hastanesi, Istanbul
- United Kingdom (4):
  - The Royal Free Hospital NHS Foundation Trust, Barnet, England
  - Royal Free London NHS Foundation Trust, London, England
  - The Christie NHS Foundation Trust, Manchester, England
  - Nottingham University Hospitals NHS Trust, Nottingham, England

IPD SHARING:
Plan to Share IPD: No